CLINICAL TRIAL: NCT07137507
Title: Comparison of Lung Expansion After Uniportal and Multiportal Video Assisted Thoracic Surgery for Stage II Post Pneumonic Bacterial Empyema Thoracis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Zeeshan Sarwar, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB/2021/873/SIMS
Record Dates: First submitted 2025-08-12; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Empyema, Pleural; Thoracic Empyema
Keywords: empyema thoracis; uniportal VATS; Multiportal VATS; Decortication; thoracotomy
MeSH Terms: conditions — Empyema, Pleural; Empyema

STUDY DESIGN:
Intervention Model Description: This study was designed as a parallel-arm randomized controlled trial to compare the effectiveness of uniportal versus multiportal video-assisted thoracic surgery (VATS) in achieving postoperative lung expansion in patients with stage II empyema
Who Masked: Investigator
Masking Description: Allocation concealment was maintained using sealed, opaque envelopes prepared by an independent staff member not involved in patient recruitment or data collection. Blinding was applied at the outcome assessment stage, with the radiologists evaluating postoperative lung expansion unaware of the surgical approach used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Uniportal Group (Experimental): Uniportal Video Assisted Thoracic Surgery group
  Interventions: Procedure: Uniportal VATS
- Multiportal Group (Experimental): Multi-portal Video Assisted Thoracic Surgery group
  Interventions: Procedure: Multi-portal VATS

INTERVENTIONS:
Procedure: Uniportal VATS — Decortication of pleural empyema is done using single-port VATS
  Arms: Uniportal Group
Procedure: Multi-portal VATS — Decortication of pleural empyema is done using two or more ports with VATS
  Arms: Multiportal Group

SUMMARY:
It was a parallel-armed randomized control study in which 160 participants admitted to the Thoracic Surgery Department, Services Hospital, Lahore were included. The participants were divided into two equal groups (80 in each group). Uniportal Group participants underwent uniportal video assisted thoracic surgery (VATS), while multiportal Group participants were treated with multiportal video assisted thoracic surgery(VATS). Simple consecutive sampling was carried out. Expansion of lung was evaluated postoperatively at the 1st, 3rd, 7th and 15th postoperative day by chest radiograph after uniportal and multiportal VATS.

DETAILED DESCRIPTION:
Empyema is a problem that thoracic surgeons deal in everyday practice. The main goal of treatment is evacuating the pus and fibrin deposits in the thoracic cavity for complete lung expansion. Traditionally, the surgical approach was open thoracotomy; then the multiportal video assisted thoracic surgery (VATS) approach became more common. Recently, more surgeons are adopting the uniportal VATS approach, which has become a powerful surgical tool, for the treatment of stage II empyema.

Uniportal and multiportal VATS are a feasible technique in all patients with pleural empyema requiring surgery. In this study, the investigators observed comparable postoperative success rates, no need for conversion, and successful completion of decortication via both multiportal and uniportal approaches. This transition to a single-incision technique was associated with fewer chest tubes, minimal surgical trauma, and no compromise in clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage II empyema
* More than 18 years old patients deemed fit for intervention.
* Both genders
* Unintubated patients

Exclusion Criteria:

* Patients with stages I and III empyema
* Patient with TB empyema
* Patient with Fungal empyema
* Patients unfit for general anesthesia.
* Unwilling to participate

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
complete lung expansion after decortication | 15 days
  Complete expansion of lung after Uniportal or Multiportal VATS was defined as, no residual pneumothorax or fluid collection on the chest radiograph, post - operatively. Lung expansion after surgery will be measured in percentages by calculating percentage of residual pneumothorax or fluid collection and was assessed using chest X-ray. Chest x-rays were performed on post-operative day 1, 3, 7 and 15. Physiologically normal and completely expanded lung is the set parameter for checking and comparing the expansion of operated lung after decortication.

SECONDARY OUTCOMES:
post-operative thoracotomy site pain | 07 days
  Recording of post-operative thoracotomy pain at the site of uniportal or multiportal VATS was also assessed on post-operative day 1, 3 and 7. The Visual Analogue Scale (VAS) is a simple, widely used tool for measuring pain intensity. It consists of a straight line, usually 10 cm in length, with two endpoints:
  "0" = no pain "10" (or 100) = worst imaginable pain The patient marks a point on the line that best represents their perceived pain level. The score is then measured in millimeters or centimeters from the "no pain" end, giving a numerical value for pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Shoaib Nabi, Study Chair — SIMS, Services Hospital, Lahore
Locations (1):
- Services Institute Of Medical Sciences, Services Hospital, Lahore, Punjab Province, Pakistan